CLINICAL TRIAL: NCT00150774
Title: A Double-blind, Multicenter, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Levetiracetam (LEV) (Oral Tablets of 500 mg b.i.d.) at a Dose of 3000 mg/Day as Adjunctive Treatment in Adolescents (≥ 12 Years) and Adults (≤ 65 Years) Suffering From Idiopathic Generalized Epilepsy With Myoclonic Seizures.
Brief Title: Levetiracetam as add-on Treatment of Myoclonic Jerks in Adolescents + Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N166
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2010-02

CONDITIONS: Generalized Convulsive Epilepsy
Keywords: Idiopathic Generalized Epilepsy, Myoclonic seizures; Keppra - Levetiracetam
MeSH Terms: conditions — Epilepsy, Generalized; Epilepsy, Idiopathic Generalized; Seizures | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
A double-blind, placebo-controlled study to assess the efficacy of adjunctive treatment with LEV 3000mg/day in reducing myoclonic seizures in adolescents and adults suffering from idiopathic generalised epilepsy and to evaluate the safety of LEV in the same population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed diagnosis consistent with idiopathic generalized epilepsy experiencing myoclonic seizures (IIB) that are classifiable according to the International Classification of Epileptic Seizures. To ensure an idiopathic generalized epilepsy population, only these subjects with the diagnosis of juvenile myoclonic epilepsy (JME), juvenile absence epilepsy (JAE) or epilepsy with generalized tonic- clonic seizures on awakening must be included.
* Presence of at least eight days with at least one myoclonic seizure (IIB) per day during the eight weeks of the Baseline period.
* Absence of brain lesion documented on a CT scan or MRI; if a CT scan or MRI has not been performed within the past five years before Visit 1, a CT scan (or MRI where legally required) should be performed during the Baseline period.
* Presence of EEG features consistent with idiopathic generalized epilepsy on an EEG recorded during the Baseline period or no more than one year before Visit 1.
* Male/female children ≥ 12 years of age or adult ≤ 65 years of age at Visit 1.
* Subject on a stable dose of one standard anti-epileptic treatment for at least four weeks before Visit 1.

Exclusion Criteria:

* Previous exposure to levetiracetam.
* History of partial seizures.
* History of convulsive or non-convulsive status epilepticus within 3 months prior to Visit 1.
* Subject taking vigabatrin or tiagabine, subject on felbamate with less than 18 months exposure, and subject under vagal nerve stimulation or ketogenic diet.
* Subject taking any drug (except the concomitant AEDs) with possible CNS effects.

Ages: 12 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 116
Dates: Start 2001-11; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Responder rate in myoclonic (type IIB) seizures days over 16 weeks

SECONDARY OUTCOMES:
Safety and tolerability of levetiracetam by means of AE, laboratory assessments, plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Rosenfeld WE, Benbadis S, Edrich P, Tassinari CA, Hirsch E. Levetiracetam as add-on therapy for idiopathic generalized epilepsy syndromes with onset during adolescence: analysis of two randomized, double-blind, placebo-controlled studies. Epilepsy Res. 2009 Jul;85(1):72-80. doi: 10.1016/j.eplepsyres.2009.02.016. Epub 2009 Mar 26. PMID 19327967
- [Result] Noachtar S, Andermann E, Meyvisch P, Andermann F, Gough WB, Schiemann-Delgado J; N166 Levetiracetam Study Group. Levetiracetam for the treatment of idiopathic generalized epilepsy with myoclonic seizures. Neurology. 2008 Feb 19;70(8):607-16. doi: 10.1212/01.wnl.0000297512.18364.40. PMID 18285535